CLINICAL TRIAL: NCT00829608
Title: Investigator Initiated Study of Effects of Progression of Recurrent Respiratory Papillomatosis in Patients After They Are Given Human Papillomavirus Quadrivalent Vaccine
Brief Title: Therapeutic Treatment With Human Papillomavirus Quadrivalent Vaccine for Recurrent Respiratory Papillomatosis
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: investigator has left the institution
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1124197
Record Dates: First submitted 2009-01-05; First posted 2009-01-27 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Recurrent Respiratory Papillomatosis
Keywords: RRP; Recurrent Respiratory Papillomatosis; HPV vaccine; HPV
MeSH Terms: conditions — Recurrent respiratory papillomatosis | interventions — Papillomavirus Vaccines; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Human Papillomavirus Vaccine (Experimental): There are 9 participants currently being followed in the faculty sponsor's clinic that carry the clinical and histologic diagnosis of RRP. The 9 participants meet one or more of the following criteria: Surgery requirement of more than 4 procedures per year, distal multisite spread of disease, and rapid regrowth of papilloma disease with airway compromise.
  Interventions: Biological: Human Papillomavirus Vaccine

INTERVENTIONS:
Biological: Human Papillomavirus Vaccine — 0.5 mL of quadrivalent HPV vaccine will be given intramuscularly at three separate intervals. Dose 2 is given 2 weeks after dose 1 and dose 3 is given 4 weeks after dose 1 for a total of 3 doses over 2 months.
  Other Names: Gardasil, HPV vaccine

SUMMARY:
The purpose of this study is to determine if administration of the HPV quadrivalent vaccine in patients diagnosed with RRP has a therapeutic effect on their clinical course. More specifically, does administration of the vaccine decrease the size and number of papillomas, severity of disease (i.e. hoarseness, inspiratory vs. biphasic stridor, airway obstruction) using the LCAS and time interval between required surgical debulking will be analyzed.

DETAILED DESCRIPTION:
Patients who carry the diagnosis of Recurrent Respiratory Papillomatosis (RRP) will be asked to participate in the study. These patients have been followed by the faculty investigator for several years. Their disease state requires frequent interventions aimed at decreasing the severity and symptomatology of their vocal fold papillomas. Patients will be given the human papillomavirus quadrivalent vaccine and their clinical course will be followed over the next 6 months. Patients will have a laryngoscopic examination prior to treatment to establish their baseline disease state. They will have repeat laryngoscopic examinations at the time of the first, second and third vaccine injections, which will be given 1 month intervals for a total of 3 doses. They will have physical exam and laryngoscopic examinations at 1 month intervals for the first 6 months after administration of the vaccine. The severity of their clinical disease will be objectively measured using a validated scale for RRP assessment, the Laryngoscopic and Clinical Assessment Scale (LCAS).

ELIGIBILITY:
Inclusion Criteria:

* There are 9 participants currently being followed in the faculty sponsor's clinic that carry the clinical and histologic diagnosis of RRP. The 9 participants meet one or more of the following criteria: Surgery requirement of more than 4 procedures per year, distal multisite spread of disease, and rapid regrowth of papilloma disease with airway compromise.

Exclusion Criteria:

* If any of the 9 patients meet the following criteria they will be excluded from the study:

  * Pregnancy
  * Hypersensitivity or allergy to vaccine components (i.e. Saccharomyces cerevisiae yeast)
  * Immunocompromised patients (i.e. patients with HIV, cancer, or who take immunosuppressant medications including all forms of steroids)
  * Have a fever over 100°F (37.8°C)
  * Moderate or severe acute illness (with or without fever)
  * Coagulopathies
  * Platelet counts of less than 100,000
  * Any history of recent treatment(within 3 months) with any investigational drug or other adjuvant RRP therapy (including interferon-gamma, ribavirin, acyclovir, cidofovir and photodynamic therapy, indole-3-carbinol)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of the pre-vaccine and post-vaccine RRP scoring assessments, intersurgical intervals, and annualized surgical rates. | 12 months

SECONDARY OUTCOMES:
The secondary end points will include changes in the RRP scoring assessment, intersurgical intervals and changes in annualized surgical rates. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Troy D Scheidt, MD, Principal Investigator — University of Missour-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No